CLINICAL TRIAL: NCT04369976
Title: Estimating the Optimal G Level for Training and Rehabilitation on a Short Arm Human Centrifuge
Brief Title: Short Arm Human Centrifuge Therapeutic Training and Rehabilitation (GRACER1)
Acronym: GRACER1
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Greek Aerospace Medical Association and Space Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 001955
Record Dates: First submitted 2020-04-15; First posted 2020-04-30 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis; Stroke; Pulmonary Disease, Chronic Obstructive; Aged
MeSH Terms: conditions — Multiple Sclerosis; Stroke; Pulmonary Disease, Chronic Obstructive | interventions — Exercise Therapy; Rehabilitation

STUDY DESIGN:
Intervention Model Description: The use of a short arm human centrifuge intervention program (SAHC) combined with exercise, compared to a standard of care (SOC) rehabilitation program in physically impaired patients with MS, stroke, severe Chronic Obstructive Pulmonary Disease (COPD) and elderly people with balance and gait disorders (risk of falls). The patients will be randomly assigned to the centrifuge training (SAHC intervention), SOC training or a passive control group. The SAHC intervention consists of 3 sessions per week. The session duration is 1 hour. The intervention will last for 3 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHORT ARM HUMAN CENTRIFUGE (Experimental): SHORT ARM HUMAN CENTRIFUGE IN COMBINATION WITH EXERCISE INTERMITTENT CENTRIFUGATION TOTAL TIME 30 MINUTES
  Interventions: Device: ARTIFICIAL GRAVITY COMBINED WITH EXERCISE

INTERVENTIONS:
Device: ARTIFICIAL GRAVITY COMBINED WITH EXERCISE — The passive control group will abstain from any exercise. Recordings of the participant's will include cardiovascular functioning cardiac output (CO), stroke volume (SV) mean arterial pressure (MAP) diastolic blood pressure (DBP), systolic blood pressure (SBP), and heart rate (HR), Electroencephalography ( EEG) as well as dynamic force and stance and muscle oxygenation. More specifically, after 6 training sessions (2 weeks), the centrifugation load will be increased and will be combined with either aerobic exercise (through an ergometer) or resistance training through elastic training bands. Functional connectivity and cortical-network features will be used by deep learning algorithms in order to define the optimal centrifuge training .
  Other Names: standard of care (SOC) rehabilitation program

SUMMARY:
The study is a single blind randomized controlled trial (RCT) designed to examine the benefit of a short arm human centrifuge intervention program (SAHC) combined with exercise, compared to a standard of care (SOC) rehabilitation program in physically impaired patients with MS, stroke, severe chronic obstructive pulmonary disease (COPD) and elderly people with balance and gait disorders (risk of falls).

DETAILED DESCRIPTION:
The patients will be randomly assigned to the short arm human centrifuge training (SAHC intervention), standard of care (SOC training) or a passive control. The SAHC intervention consists of 3 sessions per week. The session duration is 1 hour. The intervention will last 3 months.

Aiming to estimate the minimum number of participants required for obtaining reliable results, the investigators performed power analysis. It was conducted in g-power 3.1 to determine a sufficient sample size using an alpha of 0.05, a power of 0.80, and a medium effect size (f = 0.21). Based on the aforementioned assumptions, a total sample size of 26 participants per group was computed.

The passive control group will abstain from any exercise. Initially, there will be one session serving as an evaluation and familiarization of the SAHC group participants on the centrifuge. Its aim besides familiarization will be also to individually assess the optimal according to the participant's cardiovascular functioning with cardiac output (CO), stroke volume (SV) mean arterial pressure (MAP) diastolic blood pressure (DBP), systolic blood pressure (SBP), and heart rate (HR). These criteria are monitored at each training session and are used to dynamically adapt the intervention intensity. More specifically, after 6 training sessions (2 weeks), the centrifugation load will be increased and considering the cardiovascular criteria, centrifugation will be combined with either aerobic exercise (through an ergometer) or resistance training through elastic training bands. Further verification of the dynamic configuration of the intervention will be provided by the electroencephalographic (EEG) assessment. More specifically, resting state EEG (eyes open & closed condition, lying in horizontal position) and centrifugation in three different intensities, mild (corresponding to 0.5,0.7, and 1 g), medium (corresponding to 1.2 and 1.5 g) and high intensity (corresponding to 1.7 and 2 g). Functional connectivity and cortical-network features derived from graph theory will be used by deep learning algorithms (convolutional neural networks) in order to define the optimal centrifuge training.

A set of core outcomes as described below will be collected at the following experimental time instances: a) baseline, b) after 4 weeks, c) 8 weeks, d) 3 months, e) 6-month follow-up, g) 12-month follow-up. The outcomes will be collected across the domains of body structure and function, activity, and participation as classified by the world health organization international classification of functioning (ICF), disability and health.

The primary outcomes are the following:

1. A set of cardiovascular biosignal sensors described above,
2. Electroencephalographic (EEG) recordings,
3. The functional gait assessment (FGA) and
4. The functioning differences assessed by changes in summary ordinal score on the short physical performance battery (SPPB). The battery consists of three tests: balance, gait ability and leg strength. The score for each test is given in categorical modality (0-4) based on run time intervals, and the total score will range from 0 (worst) to 12 points (best). The SPPB has been shown to be a valid instrument for screening frailty and predicting disability, institutionalization and mortality. A total score of less than 10 points indicates frailty and a high risk of disability and falls. 1 point change in the total score has demonstrated to be of clinical relevance.

More primary outcomes include other measures of gaze and postural stability, fatigue, and functional mobility, isokinetic strength and muscle oxygen consumption. Additionally, a set of biomarkers in blood and urine will be collected.

ELIGIBILITY:
Inclusion Criteria:

* both male and female
* height less than 2 m,
* healthy or
* with gait disorder or
* impaired mobility from multiple sclerosis or
* stroke,
* chronic obstructive pulmonary disease (COPD) or
* elderly

Exclusion Criteria:

* Neurological or psychiatric disorder,
* vertigo,
* nausea or
* chronic pain,
* participants with a height greater than 2 meters,
* participants with chronic use of substances or alcoholism,
* with recent (within 6 months) surgery,
* current arrhythmia,
* severe migraines,
* pregnancy,
* epilepsy,
* cholelithiasis or
* kidney stones,
* dehydration,
* recent wounds from surgery,
* recent fractures (unless recommended by a doctor),
* acute inflammation or
* pain and
* newly inserted metal pins or plates, newly implanted stents .

Ages: 17 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular physiological parameter 1 cardiac output (CO) 1-standing | The time frame will include: changes from baseline up to 6 months
  Cardiac output (CO) unit L/min, measured by a non invasive tensortip device attached to the subject's finger after 5 minutes standing condition
Cardiovascular physiological parameter 1 cardiac output (CO) 2-lying | The time frame will include: changes from baseline up to 6 months
  Cardiac output (CO) unit L/min, measured by a non invasive tensortip device attached to the subject's finger after 5 minutes lying condition
Cardiovascular physiological parameter 1 cardiac output (CO) 3-mild intensity | The time frame will include: changes from baseline up to 6 months
  Cardiac output (CO) unit L/min, measured by a non invasive tensortip device attached to the subject's finger after 5 minutes mild intensity centrifugation condition
Cardiovascular physiological parameter 1 cardiac output (CO) 4-medium intensity | The time frame will include: changes from baseline up to 6 months
  Cardiac output (CO) unit L/min, measured by a non invasive tensortip device attached to the subject's finger after 5 minutes medium intensity centrifugation condition
Cardiovascular physiological parameter 1 cardiac output (CO) 5-high intensity | The time frame will include: changes from baseline up to 6 months
  Cardiac output (CO) unit L/min, measured by a non invasive tensortip device attached to the subject's finger after 5 minutes high intensity centrifugation condition
Cardiovascular physiological parameter 2, Stroke volume (SV) 1-standing | The time frame will include: changes from baseline up to 6 months
  Stroke volume (SV) unit L/beat, measured by a non invasive tensortip device attached to the subject's finger after 5 minutes standing position
Cardiovascular physiological parameter 2, Stroke volume (SV) 2-lying | The time frame will include: changes from baseline up to 6 months
  Stroke volume (SV) unit L/beat, measured by a non invasive tensortip device attached to the subject's finger after 5 minutes lying position
Cardiovascular physiological parameter 2, Stroke volume (SV) 3-mild intensity | The time frame will include: changes from baseline up to 6 months
  Stroke volume (SV) unit L/beat, measured by a non invasive tensortip device attached to the subject's finger after 5 minutes centrifugation of mild intensity (from 0,5 g to 1 g
Cardiovascular physiological parameter 2, Stroke volume (SV) 4-medium intensity | The time frame will include: changes from baseline up to 6 months
  Stroke volume (SV) unit L/beat, measured by a non invasive tensortip device attached to the subject's finger after 5 minutes centrifugation of medium intensity (from 1,2g to1,5 g
Cardiovascular physiological parameter 2, Stroke volume (SV) 5-high intensity | The time frame will include: changes from baseline up to 6 months
  Stroke volume (SV) unit L/beat, measured by a non invasive tensortip device attached to the subject's finger after 5 minutes centrifugation of high intensity (from 1,7g to 2 g)
Cardiovascular physiological parameter 3, mean arterial pressure (MAP) 1-standing | The time frame will include: changes from baseline up to 6 months
  Mean arterial pressure (MAP) unit mmHg, measured by a non invasive tensortip device attached to the subject's finger at standing position
Cardiovascular physiological parameter 3, mean arterial pressure (MAP) 2-lying | The time frame will include: changes from baseline up to 6 months
  Mean arterial pressure (MAP) unit mmHg, measured by a non invasive tensortip device attached to the subject's finger at lying position
Cardiovascular physiological parameter 3, mean arterial pressure (MAP) 3-mild intensity | The time frame will include: changes from baseline up to 6 months
  Mean arterial pressure (MAP) unit mmHg, measured by a non invasive tensortip device attached to the subject's finger after centrifugation with mild intensity (from 0,5 g to 1 g)
Cardiovascular physiological parameter 3, mean arterial pressure (MAP) 4-medium intensity | The time frame will include: changes from baseline up to 6 months
  Mean arterial pressure (MAP) unit mmHg, measured by a non invasive tensortip device attached to the subject's finger after centrifugation with medium intensity (from 1,2g to1,5 g)
Cardiovascular physiological parameter 3, mean arterial pressure (MAP) 5-high intensity | The time frame will include: changes from baseline up to 6 months
  Mean arterial pressure (MAP) unit mmHg, measured by a non invasive tensortip device attached to the subject's finger after centrifugation with high intensity (from 1,7g to 2 g).
Cardiovascular physiological parameter 4, diastolic blood pressure (DBP) 1-standing | The time frame will include: changes from baseline up to 6 months
  Diastolic blood pressure (DBP) unit mmHg,measured by a non invasive tensortip device attached to the subject's finger after 5 minutes standing position
Cardiovascular physiological parameter 4, diastolic blood pressure (DBP) 2-lying | The time frame will include: changes from baseline up to 6 months
  Diastolic blood pressure (DBP) unit mmHg,measured by a non invasive tensortip device attached to the subject's finger after 5 minutes lying position
Cardiovascular physiological parameter 4, diastolic blood pressure (DBP) 3-low intensity | The time frame will include: changes from baseline up to 6 months
  Diastolic blood pressure (DBP) unit mmHg,measured by a non invasive tensortip device attached to the subject's finger after centrifugation of mild intensity (from 0,5 g to 1 g).
Cardiovascular physiological parameter 4, diastolic blood pressure (DBP) 4-medium intensity | The time frame will include: changes from baseline up to 6 months
  Diastolic blood pressure (DBP) unit mmHg,measured by a non invasive tensortip device attached to the subject's finger after centrifugation with medium intensity (from 1,2g to1,5 g).
Cardiovascular physiological parameter 4, diastolic blood pressure (DBP) 5-high intensity | The time frame will include: changes from baseline up to 6 months
  Diastolic blood pressure (DBP) unit mmHg,measured by a non invasive tensortip device attached to the subject's finger after centrifugation of high intensity (from 1,7g to 2 g).
Cardiovascular physiological parameter 5, systolic blood pressure (SBP) 1-standing | The time frame will include: changes from baseline up to 6 months
  Systolic blood pressure (SBP) unit mmHg, measured by a non invasive tensortip device attached to the subject's finger after 5 minutes at standing position
Cardiovascular physiological parameter 5, systolic blood pressure (SBP) 2;lying | The time frame will include: changes from baseline up to 6 months
  Systolic blood pressure (SBP) unit mmHg, measured by a non invasive tensortip device attached to the subject's finger after 5 minutes at lying position
Cardiovascular physiological parameter 5, systolic blood pressure (SBP) 3-mild intensity | The time frame will include: changes from baseline up to 6 months
  Systolic blood pressure (SBP) unit mmHg, measured by a non invasive tensortip device attached to the subject's finger after 5 minutes centrifugation with mild intensity (from 0,5 g to 1 g).
Cardiovascular physiological parameter 5, systolic blood pressure (SBP) 4-medium intensity | The time frame will include: changes from baseline up to 6 months
  Systolic blood pressure (SBP) unit mmHg, measured by a non invasive tensortip device attached to the subject's finger after 5 minutes centrifugation with medium intensity (from 1,2g to1,5 g)
Cardiovascular physiological parameter 5, systolic blood pressure (SBP) 5-high intensity | The time frame will include: changes from baseline up to 6 months
  Systolic blood pressure (SBP) unit mmHg, measured by a non invasive tensortip device attached to the subject's finger after 5 minutes centrifugation with high intensity (from 1,7g to 2 g)
Cardiovascular physiological parameter 6, heart rate (HR) 1-standing | The time frame will include: changes from baseline up to 6 months
  Heart rate (HR) unit beats/min, measured by a non invasive tensortip device attached to the subject's finger after 5 minutes at standing position
Cardiovascular physiological parameter 6, heart rate (HR) 2-lying | The time frame will include: changes from baseline up to 6 months
  Heart rate (HR) unit beats/min, measured by a non invasive tensortip device attached to the subject's finger after 5 minutes at lying position
Cardiovascular physiological parameter 6, heart rate (HR) 3-mild intensity | The time frame will include: changes from baseline up to 6 months
  Heart rate (HR) unit beats/min, measured by a non invasive tensortip device attached to the subject's finger after 5 minutes centrifugation of mild intensity (from 0,5 g to 1 g).
Cardiovascular physiological parameter 6, heart rate (HR) 4-medium intensity | The time frame will include: changes from baseline up to 6 months
  Heart rate (HR) unit beats/min, measured by a non invasive tensortip device attached to the subject's finger after 5 minutes centrifugation with medium intensity (from 1,2g to1,5 g).
Cardiovascular physiological parameter 6, heart rate (HR) 5-high intensity | The time frame will include: changes from baseline up to 6 months
  Heart rate (HR) unit beats/min, measured by a non invasive tensortip device attached to the subject's finger after 5 minutes centrifugation of high intensity (from 1,7g to 2 g).
Electrical activity of the brain in alpha band, Electroencephalography (EEG)(μV) 1 | The time frame will include: changes from baseline up to 6 months
  Recording of the brain's spontaneous electrical activity using multiple electrodes placed on the scalp with a conductive gel or paste, usually after preparing the scalp area by light abrasion to reduce impedance due to dead skin cells. Electrode locations and names are specified by the International 10-20 system.Each electrode is connected to one input of a differential amplifier, which amplifies the voltage between the active electrode and the reference (typically 1,000-100,000 times, or 60-100 dB of voltage gain) and the amplified signal is digitized via an analog-to-digital converter, after being passed through an anti-aliasing filter. Analog-to-digital sampling typically occurs at 256-512 Hz in clinical scalp EEG; sampling rates of up to 20 kHz will be used .
  The recording involves the subject with eyes open.
Electrical activity of the brain in alpha band, Electroencephalography (EEG)(μV) 2 | The time frame will include: changes from baseline up to 6 months
  Recording of the brain's spontaneous electrical activity using multiple electrodes placed on the scalp with a conductive gel or paste, usually after preparing the scalp area by light abrasion to reduce impedance due to dead skin cells. Electrode locations and names are specified by the International 10-20 system.Each electrode is connected to one input of a differential amplifier, which amplifies the voltage between the active electrode and the reference (typically 1,000-100,000 times, or 60-100 dB of voltage gain) and the amplified signal is digitized via an analog-to-digital converter, after being passed through an anti-aliasing filter. Analog-to-digital sampling typically occurs at 256-512 Hz in clinical scalp EEG; sampling rates of up to 20 kHz will be used .
  The recording involves the subject with eyes closed.
Electrical activity of the brain in alpha band, Electroencephalography (EEG)(μV) 3 | The time frame will include: changes from baseline up to 6 months
  Recording of the brain's spontaneous electrical activity using multiple electrodes placed on the scalp with a conductive gel or paste, usually after preparing the scalp area by light abrasion to reduce impedance due to dead skin cells. Electrode locations and names are specified by the International 10-20 system.Each electrode is connected to one input of a differential amplifier, which amplifies the voltage between the active electrode and the reference (typically 1,000-100,000 times, or 60-100 dB of voltage gain) and the amplified signal is digitized via an analog-to-digital converter, after being passed through an anti-aliasing filter. Analog-to-digital sampling typically occurs at 256-512 Hz in clinical scalp EEG; sampling rates of up to 20 kHz will be used .
  The recording involves the subject in standing position.
Electrical activity of the brain in alpha band, Electroencephalography (EEG)(μV) 4 | The time frame will include: changes from baseline up to 6 months
  Recording of the brain's spontaneous electrical activity using multiple electrodes placed on the scalp with a conductive gel or paste, usually after preparing the scalp area by light abrasion to reduce impedance due to dead skin cells. Electrode locations and names are specified by the International 10-20 system.Each electrode is connected to one input of a differential amplifier, which amplifies the voltage between the active electrode and the reference (typically 1,000-100,000 times, or 60-100 dB of voltage gain) and the amplified signal is digitized via an analog-to-digital converter, after being passed through an anti-aliasing filter. Analog-to-digital sampling typically occurs at 256-512 Hz in clinical scalp EEG; sampling rates of up to 20 kHz will be used .
  The recording involves the subject in lying position.
Electrical activity of the brain in alpha band, Electroencephalography (EEG)(μV) 5 | The time frame will include: changes from baseline up to 6 months
  Recording of the brain's spontaneous electrical activity using multiple electrodes placed on the scalp with a conductive gel or paste, usually after preparing the scalp area by light abrasion to reduce impedance due to dead skin cells. Electrode locations and names are specified by the International 10-20 system.Each electrode is connected to one input of a differential amplifier, which amplifies the voltage between the active electrode and the reference (typically 1,000-100,000 times, or 60-100 dB of voltage gain) and the amplified signal is digitized via an analog-to-digital converter, after being passed through an anti-aliasing filter. Analog-to-digital sampling typically occurs at 256-512 Hz in clinical scalp EEG; sampling rates of up to 20 kHz will be used .
  The recording involves the subject in centrifugation with mild intensity (from 0,5 g to 1 g).
Electrical activity of the brain in alpha band, Electroencephalography (EEG)(μV) 6 | The time frame will include: changes from baseline up to 6 months
  Recording of the brain's spontaneous electrical activity using multiple electrodes placed on the scalp with a conductive gel or paste, usually after preparing the scalp area by light abrasion to reduce impedance due to dead skin cells. Electrode locations and names are specified by the International 10-20 system.Each electrode is connected to one input of a differential amplifier, which amplifies the voltage between the active electrode and the reference (typically 1,000-100,000 times, or 60-100 dB of voltage gain) and the amplified signal is digitized via an analog-to-digital converter, after being passed through an anti-aliasing filter. Analog-to-digital sampling typically occurs at 256-512 Hz in clinical scalp EEG; sampling rates of up to 20 kHz will be used .
  The recording involves the subject in centrifugation with medium intensity (from 1,2g to1,5 g).
Electrical activity of the brain in alpha band, Electroencephalography (EEG)(μV) 7 | The time frame will include: changes from baseline up to 6 months
  Recording of the brain's spontaneous electrical activity using multiple electrodes placed on the scalp with a conductive gel or paste, usually after preparing the scalp area by light abrasion to reduce impedance due to dead skin cells. Electrode locations and names are specified by the International 10-20 system.Each electrode is connected to one input of a differential amplifier, which amplifies the voltage between the active electrode and the reference (typically 1,000-100,000 times, or 60-100 dB of voltage gain) and the amplified signal is digitized via an analog-to-digital converter, after being passed through an anti-aliasing filter. Analog-to-digital sampling typically occurs at 256-512 Hz in clinical scalp EEG; sampling rates of up to 20 kHz will be used .
  The recording involves the subject in centrifugation of high intensity (from 1,7g to 2 g).
The Short Physical Performance Battery assessment score | The time frame will include: changes from baseline up to 6 months
  The functioning differences assessed by changes in summary ordinal score on Balance, gait ability and leg strength.
  The score for each test is given in categorical modality (0-4) based on run time intervals, and the total score will range from 0 (worst) to 12 points (best).
The Functional Gait Assessment (FGA) | changes in 3 months
  questionnaire
Gastrocnemius muscle oxygenation | The time frame will include: changes in 3 months
  Oxygen saturation (SmO2 (%)) of the gastrocnemius medialis muscle measured with muscle oxygen monitor" (MOXY) placed in the gastrocnemius muscle of the dominant leg during centrifugation
Biological samples 1: CATECHOLAMINES | The time frame will include: changes in 3 months
  Unit of measurement: μmol from urine and saliva samples will be collected
Biological samples 2: ADIPONECTINE | The time frame will include: changes in 3 months
  Unit of measurement: μg/mL from serum
Biological samples 3:BDNF | The time frame will include: changes in 3 months
  Unit of measurement: ng/ml from serum
Biological samples 4:MELATONINE | The time frame will include: changes in 3 months
  Unit of measurement: pg/mL from saliva
Biological samples 5:ADENOSINE | The time frame will include: changes in 3 months
  Unit of measurement: µM from saliva
Biological samples 5:TNF-α | The time frame will include: changes in 3 months
  Unit of measurement: pg/mL from serum
Biological samples 6:IL-1β | The time frame will include: changes in 3 months
  Unit of measurement: pg/mL from serum
Biological samples 7:High-sensitivity C-reactive Protein (hs-CRP) | The time frame will include: changes in 3 months
  Unit of measurement: mg/L from serum
Biological samples 8:Total leucocyte number: | The time frame will include: changes in 3 months
  Unit of measurement: number of cells x 10^3/μL from serum
Biological samples 9:sTNF-RII | The time frame will include: changes in 3 months
  Unit of measurement: pg/ml from serum
Biological samples 10:D-creatinine | The time frame will include: changes in 3 months
  Unit of measurement: mmol/l from serum
Biological samples 11:alpha-amylase | The time frame will include: changes in 3 months
  Unit of measurement: IU, from serum
Biological samples 12:secretory immunoglobulin A (sIgA) | The time frame will include: changes in 3 months
  Unit of measurement: mg/dL, from serum
Biological samples 13: cortisol (SC) mg/dL | The time frame will include: changes in 3 months
  Unit of measurement: mg/dL, from saliva
Biological samples 14: Glucose | The time frame will include: changes in 3 months
  Unit of measurement: mg/dL, from serum
Biological samples 15: ACTH | The time frame will include: changes in 3 months
  Unit of measurement: ng/liter, from plasma
Biological samples 16: Transcortin (mg/liter) | The time frame will include: changes in 3 months
  Unit of measurement: mg/liter, from serum
Biological samples 17: Total antioxidant capacity (TAC) | The time frame will include: changes in 3 months
  Unit of measurement: mM Trolox equivalent/l , from saliva
weight in kilograms, height in meters), as appropriate, or to clarify how multiple measurements will be aggregated to arrive at one reported value (e.g., weight | changes in 3 months
  unit: Kg
Height | Day 1only
  Unit:meters
Body Mass Index | changes in 3 months
  Unit: kg/m^2).

CONTACTS AND LOCATIONS:
Overall Officials: CHRYSOULA KOURTIDOU-PAPADELI, Principal Investigator — AeMC
Locations (1):
- Euromedica-Arogi Rehabilitation Center, Thessaloniki, FW, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vernikos J. Human exploration of space: why, where, what for? Hippokratia. 2008 Aug;12 Suppl 1(Suppl 1):6-9. PMID 19048086
- [Background] Hargens AR, Bhattacharya R, Schneider SM. Space physiology VI: exercise, artificial gravity, and countermeasure development for prolonged space flight. Eur J Appl Physiol. 2013 Sep;113(9):2183-92. doi: 10.1007/s00421-012-2523-5. Epub 2012 Oct 19. PMID 23079865
- [Background] Vernikos J. Artificial gravity intermittent centrifugation as a space flight countermeasure. J Gravit Physiol. 1997 Jul;4(2):P13-6. PMID 11540676
- [Background] Frett, T., Mayrhofer, M., Schwandtner, J. et al. An Innovative Short Arm Centrifuge for Future Studies on the Effects of Artificial Gravity on the Human Body. Microgravity Sci. Technol. 26, 249-255 (2014). https://doi.org/10.1007/s12217-014-9386-9 Received: 6 December 2013 / Accepted: 29 August 2014 / Published online: 19 September 2014 © Springer Science+Business Media Dordrecht 2014
- [Background] Duda KR, Jarchow T, Young LR. Squat exercise biomechanics during short-radius centrifugation. Aviat Space Environ Med. 2012 Feb;83(2):102-10. doi: 10.3357/asem.2334.2012. PMID 22303588
- [Background] Clement GR, Bukley AP, Paloski WH. Artificial gravity as a countermeasure for mitigating physiological deconditioning during long-duration space missions. Front Syst Neurosci. 2015 Jun 17;9:92. doi: 10.3389/fnsys.2015.00092. eCollection 2015. PMID 26136665
- [Background] Martina JR, Westerhof BE, van Goudoever J, de Beaumont EM, Truijen J, Kim YS, Immink RV, Jobsis DA, Hollmann MW, Lahpor JR, de Mol BA, van Lieshout JJ. Noninvasive continuous arterial blood pressure monitoring with Nexfin(R). Anesthesiology. 2012 May;116(5):1092-103. doi: 10.1097/ALN.0b013e31824f94ed. PMID 22415387
- [Background] Penaz J. (1973). "Photoelectric measurement of blood pressure, volume and flow in the finger," in Proceedings of the Digest 10th Int Conf Med Biol Engng, (Dresden: International Federation for Medical and Biological Engineering; ), 104.
- [Background] Stenger M. B., Evans J. M., Patwardhan A. R., Moore F. B., Hinghofer-Szalkay H., Rössler A., et al. (2007). Artificial gravity training improves orthostatic tolerance in ambulatory men and women. Acta Astronaut. 60 267-272. 10.3389/fphys.2018.00716
- [Background] Trigg C. (2013). Design and Validation of a Compact Radius Centrifuge Artificial Gravity Test Platform. Ph.D. thesis, Massachusetts Institute of Technology, Cambridge.
- [Background] Yang Y, Baker M, Graf S, Larson J, Caiozzo VJ. Hypergravity resistance exercise: the use of artificial gravity as potential countermeasure to microgravity. J Appl Physiol (1985). 2007 Nov;103(5):1879-87. doi: 10.1152/japplphysiol.00772.2007. Epub 2007 Sep 13. PMID 17872403
- [Result] Chriskos P, Frantzidis CA, Gkivogkli PT, Bamidis PD, Kourtidou-Papadeli C. Automatic Sleep Staging Employing Convolutional Neural Networks and Cortical Connectivity Images. IEEE Trans Neural Netw Learn Syst. 2020 Jan;31(1):113-123. doi: 10.1109/TNNLS.2019.2899781. Epub 2019 Mar 15. PMID 30892246
- [Result] LeBlanc A, Gogia P, Schneider V, Krebs J, Schonfeld E, Evans H. Calf muscle area and strength changes after five weeks of horizontal bed rest. Am J Sports Med. 1988 Nov-Dec;16(6):624-9. doi: 10.1177/036354658801600612. PMID 3239619
- [Result] Habazettl H, Stahn A, Nitsche A, Nordine M, Pries AR, Gunga HC, Opatz O. Microvascular responses to (hyper-)gravitational stress by short-arm human centrifuge: arteriolar vasoconstriction and venous pooling. Eur J Appl Physiol. 2016 Jan;116(1):57-65. doi: 10.1007/s00421-015-3241-6. Epub 2015 Aug 18. PMID 26280651
- [Result] Diaz Artiles, A., Heldt, T., and Young, L. R. (2016). Effects of artificial gravity on the cardio vascular system: computational approach. Acta Astronaut. 126, 395-410. doi: 10.1016/j.actaastro.2016.05.005.
- [Result] Katzmarzyk PT, Church TS, Craig CL, Bouchard C. Sitting time and mortality from all causes, cardiovascular disease, and cancer. Med Sci Sports Exerc. 2009 May;41(5):998-1005. doi: 10.1249/MSS.0b013e3181930355. PMID 19346988
- [Result] Diaz-Artiles A, Heldt T, Young LR. Short-Term Cardiovascular Response to Short-Radius Centrifugation With and Without Ergometer Exercise. Front Physiol. 2018 Nov 13;9:1492. doi: 10.3389/fphys.2018.01492. eCollection 2018. PMID 30483141
- [Result] Manen O, Dussault C, Sauvet F, Montmerle-Borgdorff S. Limitations of stroke volume estimation by non-invasive blood pressure monitoring in hypergravity. PLoS One. 2015 Mar 23;10(3):e0121936. doi: 10.1371/journal.pone.0121936. eCollection 2015. PMID 25798613
- [Result] Truijen J, van Lieshout JJ, Wesselink WA, Westerhof BE. Noninvasive continuous hemodynamic monitoring. J Clin Monit Comput. 2012 Aug;26(4):267-78. doi: 10.1007/s10877-012-9375-8. Epub 2012 Jun 14. PMID 22695821
- [Result] van der Spoel AG, Voogel AJ, Folkers A, Boer C, Bouwman RA. Comparison of noninvasive continuous arterial waveform analysis (Nexfin) with transthoracic Doppler echocardiography for monitoring of cardiac output. J Clin Anesth. 2012 Jun;24(4):304-9. doi: 10.1016/j.jclinane.2011.09.008. PMID 22608585
- [Result] Verma AK, Xu D, Bruner M, Garg A, Goswami N, Blaber AP, Tavakolian K. Comparison of Autonomic Control of Blood Pressure During Standing and Artificial Gravity Induced via Short-Arm Human Centrifuge. Front Physiol. 2018 Jun 25;9:712. doi: 10.3389/fphys.2018.00712. eCollection 2018. PMID 29988521
- [Result] Wang YC, Yang CB, Wu YH, Gao Y, Lu DY, Shi F, Wei XM, Sun XQ. Artificial gravity with ergometric exercise as a countermeasure against cardiovascular deconditioning during 4 days of head-down bed rest in humans. Eur J Appl Physiol. 2011 Sep;111(9):2315-25. doi: 10.1007/s00421-011-1866-7. Epub 2011 Feb 20. PMID 21336952
- [Result] Yang CB, Zhang S, Zhang Y, Wang B, Yao YJ, Wang YC, Wu YH, Liang WB, Sun XQ. Combined short-arm centrifuge and aerobic exercise training improves cardiovascular function and physical working capacity in humans. Med Sci Monit. 2010 Dec;16(12):CR575-83. PMID 21119574